CLINICAL TRIAL: NCT04782622
Title: The Combination of Apatinib and Camerlizumab for Advanced Lung Cancer Patients
Brief Title: The Combination of Apatinib and Camerlizumab for Advanced Lung Cancer Patients With Muti-line Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: ApatPEM
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: apatinib; PD-1 inhibitor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apatinib+Camrelizumab: treated with apatinib+camrelizumab
  Interventions: Drug: Apatinib+Camrelizumab

INTERVENTIONS:
Drug: Apatinib+Camrelizumab — Apatinib 250mg po qd+Camrelizumab 200mg ivdrip q14d

SUMMARY:
The combination of Apatinib and Camrelizumab for progressed NSCLC patients with muti-line therapy : a phaseⅠB clinical study.

Brief Summary: Immunotherapy has made a major progress in Lung cancer.However, challenges such as primary and acquired resistance, small fraction of benefit population and lack of predictive and prognostic biomarkers even exist. The overall objective response rate is lower than 20% in second line-treatment and the progression-free survival (PFS) is also similar to or poorer than that of conventional second-line chemotherapy. Apatinib is a novel, orally administered, multitarget receptor tyrosine kinase inhibitor that inhibits VEGFR, PDGFR, FGFR, c-Kit, and other kinases. It functions by inhibiting tumor angiogenesis and proliferative signaling pathways. We would observe and analyze the effectiveness and safety of apatinib combined with Camrelizumab for advanced NSCLC after muti-line therapy to explore the synergistic effect of anti-angiogenic agents and immunotherapy.

DETAILED DESCRIPTION:
Enrolled patients received apatinib plus Camrelizumab treatment (apatinib, 250mg, qd; Camrelizumab, 5mg/kg, iv, d1, 21day as a cycle.)

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Lung cancer Ability to comply with protocol Aged ≥ 18 years Histologically documented NSCLC that is currently locally advanced or metastatic NSCLC Disease progression during or following at least one line treatment. Measurable disease, as defined by RECIST v1.1 ECOG performance status of 0 or 1 Life expectancy ≥ 12 weeks Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment: ANC ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility) WBC counts > 2.5 × 109/L and < 15 × 109/L Lymphocyte count ≥ 0.5 × 109/L Serum albumin ≥ 2.5 g/dL Platelet count ≥ 100 × 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility) Hemoglobin ≥ 9.0 g/dL Patients may be transfused or receive erythropoietic treatment to meet this criterion.

Liver function tests meeting one of the following criteria:

AST or ALT ≤ 2.5 × upper limit of normal (ULN), with alkaline phosphatase

≤ 2.5 × ULN or AST and ALT ≤ 1.5 × ULN in conjunction with alkaline phosphatase > 2.5 × ULN Serum bilirubin ≤ 1.5 × ULN Patients with known Gilbert's disease who have serum bilirubin level ≤ 3 × ULN may be enrolled. INR and aPTT ≤ 1.5 × ULN This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 1 week prior to randomization. Creatinine clearance ≥ 30 mL/min Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration, or Modification of Diet in Renal Disease formulas may be used for creatinine clearance calculation. Note that 24-hour urine collection is not required but is allowed.

Exclusion Criteria:

Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments Leptomeningeal disease Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures Uncontrolled hypertension Perior used anti-angiogenic agents or immune checkpoint inhibitors.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Immunotherapy has made a major progress in Lung cancer.However, challenges such as primary and acquired resistance, small fraction of benefit population and lack of predictive and prognostic biomarkers even exist. The overall objective response rate is lower than 20% in second line-treatment and the progression-free survival (PFS) is also similar to or poorer than that of conventional second-line chemotherapy. Apatinib is a novel, orally administered, multitarget receptor tyrosine kinase inhibitor that inhibits VEGFR, PDGFR, FGFR, c-Kit, and other kinases. It functions by inhibiting tumor angiogenesis and proliferative signaling pathways. We would observe and analyze the effectiveness and safety of apatinib combined with Camrelizumab for advanced NSCLC after muti-line therapy to explore the synergistic effect of anti-angiogenic agents and immunotherapy.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 03.01.2021 to 03.01.2022
  Objective response rate
Progression free survival | 03.01.2021 to 03.01.2022
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaochun Zhang, Qingdao, None Selected, China

IPD SHARING:
Plan to Share IPD: No